CLINICAL TRIAL: NCT04846218
Title: Comparison Between Agonist Trigger With HCG Luteal Phase Supplementation vs HCG Trigger With Progesterone Luteal Phase Supplementation in Antagonist Controlled HyperstimulationCycle Regarding Clinical Pregnancy Rate
Brief Title: Agonist Trigger With HCG Luteal Supplementation vs HCG Trigger With Progesterone Luteal Supplementation in Antagonist Controlled HyperstimulationCycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maii medhat nawara, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-45WE
Record Dates: First submitted 2016-12-31; First posted 2021-04-15 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Progesterone; Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): They will receive a single dose of 0.2 mg triptorelin (Decapeptyl® Ipsen Pharmaceutical Company, France) and follow up with daily 125 IU HCG injections
  Interventions: Drug: hCG; Drug: Triptorelin
- Group 2 (Active Comparator): They will receive a single dose of HCG 10000 IU was given followed by progesterone supplementation with 100mg IM (Prontogest®).
  Interventions: Drug: hCG; Drug: Progesterone

INTERVENTIONS:
Drug: hCG
Drug: Progesterone
  Other Names: Prontogest
  Arms: Group 2
Drug: Triptorelin
  Other Names: Decapeptyl
  Arms: Group 1

SUMMARY:
The aim of the current study is to compare agonist trigger and HCG luteal support vs standard HCG trigger and progesterone luteal supplementation in antagonist controlled hyperstimulation cycle as regards to clinical pregnancy rate.

DETAILED DESCRIPTION:
Prospective Interventional randomized pilotstudy on patients undergoing controlled ovarian hyperstimulation.

All patients will receive a fixed dose of 150-300 IU recombinant FSH (Gonal-F; Sereno Laboratories,Madrid, Spain) for ovarian stimulation according to age, BMI and antral follicle count (AFC).

After 6 days of stimulation, FSH will be adjusted according to ovarian response.

Premature LH surge will be prevented with 0.25 mg of a GnRH antagonist (Cetrotide; Serono International, Geneva, Switzerland) starting on day 6 when two or more follicles reach a size of 18-20 mm, trigger of ovulation will be done and followed by luteal phase support according to the protocol assigned for each group.

Group 1:

A single dose of 0.2 mg triptorelin (Decapeptyl® Ipsen Pharmaceutical Company, France) and follow up with daily 125 IU HCG injections

Group 2:

A single dose of HCG 10000 IU was given followed by progesterone supplementation with 100mg IM (Prontogest®).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 39 years.
* Body mass index between 18 and 30.
* Unexplained infertility or male factor infertility

Exclusion Criteria:

* Endocrinological disorder eg.:hyperprolactenemia, Hypo or hyper thyrodism
* More than 2 previous attemptsof IVF
* Any uterine anatomical anomaly.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2020-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 1 year
  Clinical pregnancy diagnosed by pregnancy test and ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No